CLINICAL TRIAL: NCT02229760
Title: Effect of Steady State TPV/r 500 mg/200 mg on Intracellular Concentrations of Zidovudine Triphosphate and Carbovir Triphosphate
Brief Title: Effect of Steady State TPV/r on Intracellular Concentrations of Zidovudine and Carbovir for Patients With HIV
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.109
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

ARMS (1):
- TPV/r (Tipranavir co-administered with low dose ritonavir) (Experimental)
  Interventions: Drug: Tipranavir capsules; Drug: Ritonavir capsules

INTERVENTIONS:
Drug: Tipranavir capsules
Drug: Ritonavir capsules

SUMMARY:
To determine the effect of steady-state tipranavir 500 mg/ritonavir 200 mg (TPV/r) on intracellular concentrations of zidovudine triphosphate (ZDV-TP) and carbovir triphosphate (CBV-TP) and plasma viral load

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent before study participation
2. Age >18 and <60 years
3. Female patients of child-bearing potential who use a barrier contraceptive method for at least 12 weeks before administration of study medication, during the study and for 28 days after administration of study medication has ended and who have a negative pregnancy test result
4. Ability to swallow capsules without difficulty
5. A Body Mass Index (BMI) between 18 and 29 kg/m2
6. Reasonable probability of completing the study
7. A medical history, physical examination, and electrocardiogram (ECG) before entering the study
8. Agreement to abstain from alcohol from Day -2 to Day 24
9. Agreement to abstain from ingesting grapefruit, grapefruit juice, Seville oranges or orange marmalade from Day -2 to Day 24
10. Negative urine drug screen for drugs of abuse
11. Documented HIV-1 RNA load (by PCR) at screening of <50 copies/mL for at least 3 months and on a stable ZDV or ABC regimen for at least 6 months. Acceptable documentation included laboratory data, letter, or verbal report from another provider noted in the patient's records
12. All HIV-infected patients must be TPV naïve and must not have received a PI based regimen within 6 months of enrollment

Exclusion Criteria:

1. Female patients who had a positive serum pregnancy test during the screening period of Day -14 to Day -7 or who plan to breast-feed at time (Day 0 to 30 after TPV/r administration)
2. Use of any other investigational medicine within 30 days before Day 0
3. Use of any known CYP3A4 altering drug (i.e., phenothiazines, cimetidine, barbiturates, ketoconazole, fluconazole, rifampin, steroids and herbal medications) within 30 days before Day 0. No antibiotics were permitted within 10 days before Day 0
4. Ingestion of grapefruit, grapefruit juice, Seville oranges, or orange marmalade within 2 days of study entry (Day 0)
5. Blood or plasma donations (>100 mL total) for research or altruistic reasons within 30 days before Day 0
6. Seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/minute or >90 beats/minute
7. History of any illness (including malabsorption, irregular food intake, gastrointestinal intolerance, or allergy) that, in the opinion of the investigator, might confound the results of the study or pose additional risks in administering TPV/r
8. Any acute illness within 2 weeks before Day 0
9. Patients who were currently taking any over-the-counter medication within 7 days before Day 0, or who were currently taking any prescription drug that, in the opinion of the investigator (in consultation with the BI medical monitor or pharmacokineticist), would have interfered with either the absorption, distribution, or metabolism of TPV or ritonavir
10. Hypersensitivity to TPV, ritonavir, or sulfonamide containing drugs, or antiretroviral drugs (marketed or experimental use as part of clinical research studies)
11. Sulfonamide allergy, that in the opinion of the investigator, might confound the results of the study or pose additional risks in administering TPV/r
12. Any laboratory value outside the normal reference range that is of clinical relevance at screening, according to the judgment of the investigator (i.e., aspartate aminotransferase and alanine aminotransferase levels 2.5-fold and 2.5-fold higher than the upper normal limit, respectively)
13. Based on the compliance diary, the patient had less than 100% documented compliance for 7-14 days of background Antiretroviral (ARV) (i.e., ZDV and ABC) medications before Day -5 to 0 (visit 2)
14. Use of any protease inhibitors (i.e., fosamprenavir, amprenavir, indinavir, saquinavir, lopinavir, ritonavir, atazanavir, and nelfinavir) within 6 months of enrollment
15. Patients who are co-infected with active Hepatitis B and/or C as determined by hepatitis serology.
16. Use of any anti-platelet medications (e.g. aspirin, dipyridamole, clopidogrel, or any over the counter anti-platelet medicine).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
AUC0-12h (Area under curve) of intracellular ZDV-TP | Up to 12 hours after drug administration
AUC0-12h (Area under curve) of carbovir-TP | Up to 12 hours after drug administration

SECONDARY OUTCOMES:
Number of patients with clinical significant findings in vital sings | Up to 14 days after last drug administration
Number of patients with clinical significant findings in physical examinations | Up to 14 days after last drug administration
Number of patients with clinical significant findings in laboratory measurements | Up to 14 days after last drug administration
Concentration of Zidovudine (ZDV) in plasma | Up to 14 days after drug administration
Concentration of Abacavir (ABC) in plasma | Up to 14 days after drug administration
Concentration of Tipranavir (TPV) in plasma | Up to 14 days after drug administration
Concentration of ritonavir in plasma | Up to 14 days after drug administration
Cmax (Maximum observed concentration) | Up to 14 days after drug administration
Cp12h (Trough plasma concentration) | Up to 14 days after drug administration
AUC0-12h (Area under curve) | Up to 14 days after drug administration
Number of patients with adverse events | Up to 14 days after last drug adminnistration
Percentage of patients with viral load (VL) <50 | Up to 14 days after last drug adminnistration